CLINICAL TRIAL: NCT03819231
Title: Mindfulness Training Plus Oxytocin to Reduce Smoking and Craving Among Smokers in Withdrawal
Brief Title: Mindfulness Training Plus Oxytocin Effects on Smoking Behavior
Acronym: MOXY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study completed early due to COVID-19 pandemic regulations.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, David Black, Associate Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-17-00972
Record Dates: First submitted 2019-01-16; First posted 2019-01-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Smoking; Smoking Cessation
Keywords: Mindfulness; Oxytocin
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Oxytocin; Mindfulness; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mindfulness and intranasal oxytocin (Experimental): Given oxytocin through intranasal administration and self-directed mindfulness training.
  Interventions: Drug: Oxytocin; Behavioral: Mindfulness
- Mindfulness and placebo (Active Comparator): Given sterile saline through intranasal adminstration and self-directed mindfulness training.
  Interventions: Behavioral: Mindfulness; Drug: Saline Solution
- Sham mindfulness and placebo (Sham Comparator): Given sterile saline through intranasal adminstration and sham self-directed mindfulness training.
  Interventions: Drug: Saline Solution; Behavioral: Sham mindfulness

INTERVENTIONS:
Drug: Oxytocin — A single 40 IU dose of Pitocin (oxytocin, USP; concentration = 10 IU/1 mL; PAR Pharmaceuticals, NY, USA) will be self-administered to each participant. Each 40 IU dose will be transferred into four, 1 ml intranasal atomizers and will be administered in four sprays to each nostril over the course of 15 minutes.
  Arms: Mindfulness and intranasal oxytocin
Behavioral: Mindfulness — Participants will be instructed to listen to and practice a 20-minute guided mediation each day for 7 days prior to the experimental session. The guided mindfulness practices will include body scan and seated stillness meditations.
  Arms: Mindfulness and intranasal oxytocin; Mindfulness and placebo
Drug: Saline Solution — A single 40mL doses of sterile saline (0.9% provided by USC pharmacy) will be transferred into four, 1 ml intranasal atomizers and will be self-administered in four sprays to each nostril over the course of 15 minutes.
  Arms: Mindfulness and placebo; Sham mindfulness and placebo
Behavioral: Sham mindfulness — The mindfulness sham group will be required to listen to 20-minutes of Tedtalk podcasts each day that match the attention and time of the mindfulness group. Participants will be instructed to listen to two 10-minutes segments per day in succession between lab visits while in a seated posture.
  Arms: Sham mindfulness and placebo

SUMMARY:
The purpose of this study is to examine the effects of mindfulness training and a drug called oxytocin on smoking.

DETAILED DESCRIPTION:
Mindfulness training allows individuals to be present with their own emotions, thoughts, and bodily sensations without reactive judgment, and will be given in the form of daily audio recordings. Oxytocin is a naturally occurring hormone in the brain and throughout the body. It is also an FDA-approved drug to help induce labor in pregnant women. In this study, the use oxytocin is experimental and is in the form of a nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Smoke at least 10 cigarettes per day for the past year

Exclusion Criteria:

* Current DSM-5 substance use disorder
* Any medial condition that would increase risk for study participation
* Women who are pregnant or nursing
* Current use of psychiatric medication for anxiety or mood disorders
* Planning to quit or reduce smoking in the next 30 days
* Current regular use of other nicotine-containing products
* Current mindfulness or mediation practice of greater than 5 minutes per day

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Smoking Lapse Analogue Task (delay score) | 2 hours after nasal spray administration
  This task measures ability to resist the temptation to initiate smoking under conditions in which it is advantageous to remain abstinent. The "delay score" is the number of minutes before participants begin smoking (0-50 min).
Trier Social Stress Test | 1 hour after nasal spray administration
  This test measures self-reported responses to stress in a lab setting over the course of 30 minutes through salivary cortisol and heart rate variability.

SECONDARY OUTCOMES:
Systolic blood pressure | Throughout study completion, an average of two weeks.
Diastolic blood pressure | Throughout study completion, an average of two weeks.
Heart rate | Throughout study completion, an average of two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kirkpatrick, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No